CLINICAL TRIAL: NCT01012063
Title: Perioperative Intravenous Iron With Erythropoietin for the Prevention of Postoperative Severe Anemia and Reduction of Transfusion in Bilateral Total Knee Replacement Arthroplasty
Brief Title: Perioperative Iron With Erythropoietin in Bilateral Total Knee Replacement Arthroplasty (TKRA)
Acronym: SNUBH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-0905/076-005
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Anemia; Transfusion
Keywords: iron; erythropoietin; hemoglobin; Total knee replacement arthroplasty
MeSH Terms: conditions — Anemia | interventions — Ferric Oxide, Saccharated; epoetin beta; Saline Solution; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group IE (Experimental): The group IE received iron sucrose and erythropoietin-β (Epo-β) during the operation
  Interventions: Drug: iron sucrose, erythropoietin-β
- group C (Placebo Comparator): The group C received saline as same method.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: iron sucrose, erythropoietin-β — The 200 mg of iron sucrose diluted with 100 ml of normal saline was given intravenously over one hour and the 3000 IU of Epo-β was injected subcutaneously.
  Other Names: Venoferrum; recormon
  Arms: group IE
Drug: normal saline — 100 ml of normal saline was given intravenously over one hour and 0.5ml was injected subcutaneously.
  Other Names: sodium chloride
  Arms: group C

SUMMARY:
The object of this study is to evaluate whether low dose intravenous iron and erythropoietin (Epo) can decrease transfusion requirement after the bilateral TKRA.

DETAILED DESCRIPTION:
Total knee replacement arthroplasty (TKRA) in severe osteoarthritis usually requires extensive soft tissue and bone dissection associated with substantial bleeding. Because TKRA is performed with a pneumatic tourniquet, intraoperative bleeding is not substantial, however, over 80% of the total blood loss occurs within the first 24 hour after the operation and the hidden blood loss is 50% of the total loss, making the true blood loss twice. Consequently, many patients can become anemic at early postoperative period and this anemic condition may lead to overall physical deterioration which include fatigue, dizziness, reduced exercise tolerance and delayed recovery.

Therefore, many patients frequently received the autologous or allogenic blood transfusion. In order to reduce the allogenic blood transfusion (ABT), various methods have been used, such as preoperative autologous blood donation (PABD), use of pharmacologic agents, iron or erythropoietin (Epo) and postoperative blood salvage. All of the above methods have been proved to reduce the ABT effectively6, without increase in cost.

Iron and Epo have been used widely in a variety of clinical situations instead of allogenic RBC transfusion. They also have been used for augmenting PABD or improving preoperative hemoglobin (Hb) level. However, there still remains a controversy about the efficacy of the method on the postoperative anemia. We think that these various results may be related with individual iron state of the patients and dose of drug or timing of drug application.

In this trial, iron and Epo are planned to be administered to the iron deficient non anemic patients during the operation and once again after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing bilateral total knee replacement arthroplasty
* American society of anesthesiologist class 1-3
* Hb>100 g/L
* Either serum ferritin<100 ng/ml or 100<ferritin<300 ng/ml with a transferrin saturation (TSAT) <20%

Exclusion Criteria:

* Hematologic disease
* Thromboembolic disease
* Hepatic or renal disease
* Coagulation disorder
* Infection
* Malignancy
* Under anticoagulant therapy
* Hypersensitivity to iron sucrose or Epo
* Preoperative autologous blood donation
* Use of iron or Epo and blood transfusion within the previous 1 month

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
postoperative hemoglobin | postoperative 1, 2, 3, 5 day and 2, 6 week

SECONDARY OUTCOMES:
serum iron, ferritin, total iron binding capacity (TIBC) and transferrin saturation (TSAT) | preoperation and postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Hyoseok Na, pf, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea